CLINICAL TRIAL: NCT02224352
Title: VentFree: A Novel Abdominal Stimulator to Assist With Ventilator Weaning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Collaborators: RML Specialty Hospital (Other)
Responsible Party: Principal Investigator, Franco Laghi, MD, Staff Physician, Edward Hines Jr. VA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NSF-1417104
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: COPD; Weaning Failure
Keywords: Electric Stimulation; Respiration; Abdominal wall; Lung Diseases; Respiratory Tract Diseases; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single-Arm Study (Experimental): Functional neuromuscular electrical stimulation of abdominal-wall muscles triggered by an airway pressure signal
  Interventions: Device: Functional neuromuscular electrical stimulation

INTERVENTIONS:
Device: Functional neuromuscular electrical stimulation

SUMMARY:
Background: Over one million patients in the US are estimated to undergo mechanical ventilation every year, and approximately 300,000 of them fail attempts at weaning. The morbidity and mortality of these patients is greater than in patients who are successfully weaned. It follows that treatments aimed at reducing the duration of mechanical ventilation have the potential to benefit society both in terms of human suffering and cost.

Patients who fail attempts at weaning assist their inspiratory muscles during inhalation by recruiting their expiratory muscles during exhalation. Unfortunately, this recruitment occurs relatively late during a weaning trial. The knowledge that (a) expiratory muscle recruitment can assist inspiration, (b) the recruitment of the expiratory muscles is delayed during weaning, and (c) that the respiratory muscles in patients requiring mechanical ventilation are in a catabolic state raises the possibility that strategies designed to produce an early recruitment, and improve the strength, of the expiratory muscles could improve weaning outcomes in difficult to wean patients.

The current investigation, which will be conducted in healthy subjects and in ambulatory patients with chronic obstructive pulmonary disease (COPD) at Edward Hines Jr. VAH (Aims 1 and 2), and in patients who are difficult to wean from mechanical ventilation at RML Specialty Hospital, Hinsdale, IL (Aim 3), has been designed to develop and assess a novel triggering algorithm (VentFree), that controls the delivery of non-invasive neuro muscular electrical stimulation (NMES) to the abdominal-wall muscles during exhalation, and to study the physiological (respiratory) responses to such stimulation in assisting respiration in healthy subjects, in ambulatory patients with COPD and in patients requiring pronged mechanical ventilation.

ELIGIBILITY:
Aim 1 and Aim 2:Healthy Subjects and Ambulatory COPD Patients Studied at Hines VAH

Healthy subjects (Hines VAH), Inclusion criteria:

* Age ≥ 18 years
* No history of acute or chronic respiratory disease, cardiac or neuromuscular disease.

Ambulatory COPD patients (Hines VAH), Inclusion criteria:

* Age ≥ 18 years
* Chronic airway obstruction defined as forced expiratory volume in one second (FEV1) of 70% predicted or less, ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC) of 0.7 or less
* Stable clinical condition without an exacerbation during the preceding four weeks

Aim 3: Patients being weaned from prolonged mechanical ventilation (RML Specialty Hospital), Inclusion criteria:

* Age ≥ 18 years
* History of neuromuscular disease
* Body mass index > 35 kg/m2
* Patients who have received mechanical ventilation for at least 14 days and the primary physician judges the patient is ready to start weaning
* Able to breathe spontaneously for more than 5 minutes and less than 12 hours
* Clinically stable: oxygen saturation > 90% with a fractional inspired oxygen ≤ 0.40, external PEEP ≤ 5 cm H2O, temperature ranging from 35.5 to 38.5Co, no intravenous administration of vasoactive agents.

Additional inclusion/exclusion criteria for all potential participants

* Subjects with implanted electronic devices - such as cardiac pacemakers, defibrillators and intrathecal pumps - will be excluded because NMES could cause malfunction of those devices.
* Only subjects with intact abdominal-wall skin will be enrolled because NMES can cause discomfort when applied over skin that is irritated or on open wounds.
* Pregnancy will be a contraindication to participate in the study because it is unknown whether the application of NMES to the abdominal or lumbar area during pregnancy may produce adverse effects.
* Unable to comprehend and interact in English.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-07; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 10 minutes of resting breathing
  Number of breaths that are correctly stimulated during exhalation over the total number of breaths taken.
Error rate | 10 minutes of resting breathing
  Number of false positive stimulation triggers over the total number of breaths taken.

SECONDARY OUTCOMES:
Tidal volume | 10 minutes of resting breathing
Respiratory rate | 10 minutes of resting breathing
Minute ventilation | 10 minutes of resting breathing
Esophageal pressure time product | 10 minutes of resting breathing
Trans diaphragmatic pressure time product | 10 minutes of resting breathing
Tension time index of the diaphragm | 10 minutes of resting breathing
Ratio of tidal change in Pga to tidal change in Pes | 10 minutes of resting breathing

CONTACTS AND LOCATIONS:
Overall Officials: Franco Laghi, MD, Principal Investigator — Staff Physician
Locations (2):
- United States (2):
  - Edward G. Hines Jr., VA Hospital, Hines, Illinois
  - RML Specialty Hospital, Hinsdale, Illinois